CLINICAL TRIAL: NCT06585930
Title: Study of the Relationship Between the Value of PCS (Platelet Clot Stiffness - Parameter Evaluating Platelet Participation in Clot Formation) Obtained by Sonorheometric Method of Delocalized Hemostasis (QUANTRA®), and the Presence of a Disorder of Primary Hemostasis, in Cardiac Surgery Patients. PLAQUA-Study
Brief Title: Relation Between the Value of Platelet Clot Stiffness (PCS) Obtained by Sonorheometric Method of Delocalized Hemostasis (QUANTRA®), and the Presence of a Disorder of Primary Hemostasis, in Cardiac Surgery Patients. PLAQUA-Study
Acronym: PLAQUA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A01342-45
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Primary Haemostasis Disorder in Cardiac Surgery Patients
Keywords: Primary haemostasis disorder; Platelet Clot Stiffness; QUANTRA; von Willebrand factor deficiency
MeSH Terms: conditions — Von willebrand factor, deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Blood sample — Additional 8.1 ml blood sample

SUMMARY:
The goal of this study is to determine whether the Platelet Clot Stiffness (PCS) measured by QUANTRA® is predictive of an abnormality in primary haemostasis intraoperatively in cardiac surgery performed under extracorporeal circulation.

The aim is to compare the assessment of platelet function by QUANTRA® (data called PCS, obtained in around ten minutes) with laboratory tests which are validated, but which cannot be used in current practice (response time too long, in particular). We are therefore seeking to determine whether QUANTRA is reliable in the search for a primary hemostasis anomaly, defined by significant thrombocytopenia (platelet count below 100G/L), and/or a prolongation of platelet occlusion time measured by PFA-200® (normal or increased).

This clinical research project will last 12 months. It will take place in the cardiac surgery operating room at CHU Félix Guyon, and will involve 100 patients.

Patients who have consented to participate in this research project will be managed in the operating room in the usual way, with no change to their usual care (in terms of treatments received). At the end of the surgery, we will add 3 blood samples (maximum 8.1ml) for analysis to assess platelet function and compare with QUANTRA data.

This blood sample will be the only procedure performed. Medical management remains standard and will not be disrupted by this test.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Hospitalized for scheduled cardiac surgery performed under extracorporeal circulation, including coronary bypass, valve replacement, aortic arch and combined surgeries.

Exclusion Criteria:

Patients:

* with preoperative hematocrit < 35% and preoperative platelet count < 80,000 G/L (validity of PFA-200® Test)
* With known congenital or acquired Willebrand's disease, or known platelet dysfunction.
* On double antiaggregation, not discontinued at the time of surgery
* Vulnerable patients: minors or protected adults, pregnant women, patients not affiliated to the social security system.
* Emergency situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this study were those hospitalized for scheduled cardiac surgery performed under extracorporeal circulation (including coronary bypass, valve replacement, aortic arch and combined surgeries), at the Centre Hospitalier Universiataire de la Réunion, Hopital Félix Guyon.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Presence of a primary haemostasis disorder | Two years
  Significant thrombocytopenia (platelet count below 100G/L), and/or prolonged platelet occlusion time measured by PFA-200® (normal or increased), depending on the PCS value obtained by QUANTRA®.

CONTACTS AND LOCATIONS:
Overall Officials: Margot CARON, Dr, Principal Investigator — University Hospital of Reunion Island
Locations (1):
- University Hospital of Reunion Island - Cardiac reanimation department, Saint-Denis, Réunion, Reunion

IPD SHARING:
Plan to Share IPD: No